CLINICAL TRIAL: NCT06848530
Title: Neurophysiology of the Basal Ganglia, Thalamus, and Cerebellum in Patients With Movement Disorders
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Principal Investigator, Lauren Hammer, Assistant Professor of Neurology, University of Pennsylvania
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 857558
Record Dates: First submitted 2025-02-21; First posted 2025-02-27 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-12

CONDITIONS: Movement Disorders
MeSH Terms: conditions — Movement Disorders

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Participants without Deep Brain Stimulators (Experimental): Multimodal neurophysiology (for example, electroencephalography and electromyography) will be measured during the following:
  Movement disorder medication administration -The patient's movement disorders medications, prescribed by their treating physicians outside of this study, may be administered during an experimental session.
  Interventions: Other: Prescribed Medications
- Participants with Deep Brain Stimulators (Experimental): Multimodal neurophysiology (for example, electroencephalography and electromyography) will be measured during the following:
  Movement disorder medication administration -The patient's movement disorders medications, prescribed by their treating physicians outside of this study, may be administered during an experimental session.
  Deep brain stimulator (DBS) adjustment - Participants who have had deep brain stimulation implantation as part of their standard-of-care clinical treatment may participate in this study. The patient's stimulator may be adjusted within normal clinical limits during an experimental session.
  Interventions: Other: Prescribed Medications; Other: Deep brain stimulation adjustment

INTERVENTIONS:
Other: Prescribed Medications — participant's movement disorders medications, prescribed by their treating physician
Other: Deep brain stimulation adjustment — Deep brain stimulator parameters may be adjusted within normal clinical limits
  Arms: Participants with Deep Brain Stimulators

SUMMARY:
The research study is being conducted to better understand parts of the human brain called the cortex, basal ganglia, thalamus, and cerebellum in patients with movement disorders (such as Parkinson's disease, essential tremor, dystonia, or ataxia). These brain structures are involved in movement disorders. This study attempts to better understand the brain electrical activity associated with these disorders, both in patients with and without deep brain stimulation (DBS). Recordings are made from the scalp with a noninvasive electrode and/or through the DBS stimulator if the participant has a stimulator model that is able to sense brain activity. These recordings are analyzed along with measures of movement disorder symptoms to identify brain signal signatures of symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Patients 18 years of age and above
* Any patient who has been diagnosed by a movement disorders neurologist with one of the following movement disorders:
* Parkinson's disease
* Dystonia
* Tremor, including essential tremor
* Cerebellar ataxia
* Other hyperkinetic movement disorders, such as chorea and tics

Exclusion Criteria:

- Patients with dementia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2030-04 (Estimated); Study Completion 2030-04 (Estimated)

PRIMARY OUTCOMES:
Neural signal biomarkers | 5 years
  Spatiotemporal patterns of brain neural activity (neural signal biomarkers / neurophysiologic signatures) associated with movement disorders symptoms.

CONTACTS AND LOCATIONS:
Locations (1):
- Pennsylvania Hospital, Philadelphia, Pennsylvania, United States